CLINICAL TRIAL: NCT00088751
Title: Treatment Study for Frontotemporal Dementia
Brief Title: Treatment Study of Frontotemporal Dementia
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040247; 04-N-0247
Record Dates: First submitted 2004-07-31; First posted 2004-08-02 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-06-01

CONDITIONS: Frontotemporal Lobar Degeneration
Keywords: Frontotemporal Dementia; Alzheimer's Disease; Atypical Antipsychotic; Stimulant; Apathy; Disinhibition; Antipsychotic; Biomarkers; Dementia; FTD
MeSH Terms: conditions — Frontotemporal Lobar Degeneration; Frontotemporal Dementia; Alzheimer Disease; Lethargy; Dementia

SUMMARY:
Objectives. The proposed clinical study has two goals: First, to assess the efficacy of a central nervous system stimulant and an atypical antipsychotic in treating the behavioral symptoms of FTD and second, to further characterize the biological markers, including genetic, imaging, and CSF proteins, of FTD in relation to our existing group of Alzheimer's patients.

Rationale. Frontotemporal dementia (FTD) is increasingly recognized as an important neuropsychiatric disorder. Symptoms of FTD include disinhibition, impulsivity, apathy, affective lability, and language dysfunction. The clinical syndrome is associated with frontal and/or anterior temporal atrophy on imaging and autopsy. Levels of the CSF proteins tau and (Beta)-amyloid 1-42, shown to have diagnostic utility in patients with Alzheimer's Disease (AD), have also been found to be abnormal in FTD. FTD is less associated with APOE genotype than AD, however some familial cases of FTD are associated with specific mutations in the gene encoding the tau protein. Currently, no treatments have been proven to be effective for altering the course or clinical symptoms of FTD.

Design. Study subjects will include 50 male and female patients with mild-moderate frontotemporal dementia recruited from participants in NINDS protocol 02-N-0001. In a double-blinded crossover 11-week study without a placebo control, patients will be treated with a stimulant (dextroamphetamine) and an atypical antipsychotic (quetiapine). The primary outcome measures will be the Neuropsychiatric Inventory and the Clinical Global Impression of Change. Cerebrospinal fluid, cognitive and genetic measures, brain MRIs, and side effects scales will also be collected.

DETAILED DESCRIPTION:
Objectives. The goal of the proposed clinical study is to assess the efficacy of a central nervous system stimulant and an atypical antipsychotic in treating the behavioral symptoms of FTD.

Rationale. Frontotemporal dementia (FTD) is increasingly recognized as an important neuropsychiatric disorder. Symptoms of FTD include disinhibition, impulsivity, apathy, affective lability, and language dysfunction. The clinical syndrome is associated with frontal and/or anterior temporal atrophy on imaging and autopsy. Currently, no treatments have been proven to be effective for altering the course or clinical symptoms of FTD.

Design. Study subjects will include 20 male and female patients with mild-moderate frontotemporal dementia recruited from participants in NINDS protocols 02-N-0001 and 81-N-0010. In a double-blinded crossover 11-week study without a placebo control, patients will be treated with a stimulant (dextroamphetamine) and an atypical antipsychotic (quetiapine). The primary outcome measures will be the Neuropsychiatric Inventory and the Clinical Global Impression of Change. Cognitive measures and side effects scales will also be collected.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. FTD as diagnosed by the Lund-Manchester criteria including patients with diagnoses of Semantic Dementia or Primary Progressive Aphasia.
  2. Ages 45 to 95 years old.
  3. Mild-to-moderate (CDR 1 to 2) FTD with an assigned durable power of attorney.

EXCLUSION CRITERIA:

1. Diagnosis of any form of dementia besides FTD, including AD, Lewy body dementia, vascular dementia, dementia associated with Parkinson's disease, Corticobasal Degeneration and Progressive Supranuclear Palsy.
2. Severe dementia (CDR 3).
3. Known allergy or serious adverse reaction to quetiapine or dextroamphetamine.
4. Patient is already receiving a stimulant (methylphenidate, dextroamphetamine, pemoline, or modafinil), or an antipsychotic medication, typical or atypical, including prochlorperazine and metoclopromide.
5. Patients taking any of the following medications because of their potential interaction with dextroamphetamine: MAO use currently or within 14 days prior to start of study, Furazolidone, Guanethidine, norepinephrine, sibutramine, tricyclic antidepressants, carbonic anhydrase inhibitors.
6. Patients taking the following medications because of their potential interaction with quetiapine: Carbamazepine, clozapine, lithium, thioridazine.
7. History of CVA, or at significantly increased risk for CVA (e.g., atrial fibrillation, recent TIA etc.).
8. Symptomatic cardiovascular disease (i.e., angina, claudication, TIAs, syncope), uncontrolled hyper or hypotension, or a tic disorder.
9. Any medical contraindication to performing the procedures involved in the study including blood draws or lumbar puncture.
10. We will require a woman of child-bearing age to have a pregnancy test prior to starting the study medications and to use contraception during the course of the study.
11. Patients with a previous negative trial of a stimulant.
12. Patients with a history of severe psychosis.
13. Patients with a history of recent substance abuse.
14. Patients with QTc prolongation on a baseline EKG.
15. A score of 2 or less on the Communication Functional Ratings - Swallowing Domain.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-07-23; Study Completion 2009-06-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Woods SW, Tesar GE, Murray GB, Cassem NH. Psychostimulant treatment of depressive disorders secondary to medical illness. J Clin Psychiatry. 1986 Jan;47(1):12-5. PMID 3941052
- [Background] Satel SL, Nelson JC. Stimulants in the treatment of depression: a critical overview. J Clin Psychiatry. 1989 Jul;50(7):241-9. PMID 2567730
- [Background] Galynker I, Ieronimo C, Miner C, Rosenblum J, Vilkas N, Rosenthal R. Methylphenidate treatment of negative symptoms in patients with dementia. J Neuropsychiatry Clin Neurosci. 1997 Spring;9(2):231-9. doi: 10.1176/jnp.9.2.231. PMID 9144102